CLINICAL TRIAL: NCT03722849
Title: A Functional Magnetic Resonance Imaging Study to Investigate ATP-sensitive Cough Neural Pathways in Patients With Chronic Cough Hypersensitivity
Brief Title: Functional Magnetic Resonance Imaging of ATP Cough in Chronic Cough Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stuart Mazzone (Other)
Collaborators: Imperial College London (Other); Queen's University, Belfast (Other); Monash University (Other)
Responsible Party: Sponsor-Investigator, Stuart Mazzone, Professor of Neuroscience, University of Melbourne
Organization: University of Melbourne (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Study 58136
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-03

CONDITIONS: Cough
Keywords: functional brain imaging; ATP; Capsaicin; Refractory cough
MeSH Terms: conditions — Cough | interventions — Adenosine Triphosphate; Capsaicin; Functional Neuroimaging

STUDY DESIGN:
Intervention Model Description: The experiment will consist of two sessions. The first session will involve questionnaires, followed by measures of sensitivity and behavioural responses to tussive (cough evoking) stimulation. The second session will involve functional brain imaging measures of responses to tussive stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic cough participant (Experimental): Twenty-five (25) Idiopathic chronic cough patients, defined as refractory to disease modifying therapies (eg anti-asthma medications), will be recruited.
  Participants will attend two sessions. In the first they will inhale in a single breath a nebulized solutions of increasing doses of Adenosine Triphosphate (ATP; 0.2-300 milliM) and capsaicin (0.5-125 microM) to determine their individual cough and urge-to-cough thresholds. In the second session, participants will undergo functional brain imaging (fMRI) for 1 hour while inhaling over 24 seconds randomly administered nebulized solutions of saline, or threshold doses of ATP or capsaicin.
  Interventions: Drug: Adenosine Triphosphate; Drug: Capsaicin; Other: Functional Brain Imaging
- Healthy control participant (Experimental): Twenty-five (25) appropriately age and sex matched healthy non-smoking individuals will be recruited as the comparison group.
  Participants will attend two sessions. In the first they will inhale in a single breath a nebulized solutions of increasing doses of ATP (0.2-300 milliM) and capsaicin (0.5-125 microM) to determine their individual cough and urge-to-cough thresholds. In the second session, participants will undergo fMRI for 1 hour while inhaling over 24 seconds randomly administered nebulized solutions of saline, or threshold doses of ATP or capsaicin.
  Interventions: Drug: Adenosine Triphosphate; Drug: Capsaicin; Other: Functional Brain Imaging

INTERVENTIONS:
Drug: Adenosine Triphosphate — Participants will inhale escalating concentrations of Adenosine Triphosphate (ATP) to induce cough and the urge-to-cough
  Other Names: ATP
Drug: Capsaicin — Participants will inhale escalating concentrations of capsaicin to induce cough and the urge-to-cough
Other: Functional Brain Imaging — Participants will have scans of their brain activity using 3 Tesla (3T) brainstem restricted functional brain imaging (fMRI)
  Other Names: fMRI

SUMMARY:
Persistent cough is a distressing symptom for people with respiratory disorders. Patients also often experience an ongoing urge-to-cough that prompts coughing, and which fails to resolve the sensation. Understanding how the brain controls cough and the urge-to-cough could lead to new cough suppressing therapies. The overall objective of this project is to use functional brain imaging (fMRI) to identify brain regions that are involved in the exaggerated urge-to-cough in humans with chronic cough. Our focus will be on the brainstem where information from the airways first arrives in the central nervous system.

DETAILED DESCRIPTION:
Peripheral effects of ATP via P2X3 receptors

ATP has been shown to be a tussive agent particularly on chronic cough patients who were more sensitive than non-cough subjects to inhaled ATP. ATP has been shown to augment the cough response to capsaicin in patients with asthma. Gefapixant at a single oral dose of 50 mg did not modulate capsaicin cough responses in normal volunteers and chronic cough subjects while inhibiting ATP-induced cough particularly in chronic cough subjects. These observations would suggest that ATP has a direct effect on a subset sensory neurons that evoke coughing through the activation of P2X3 receptors.

The use of fMRI to provide insights into the peripheral and central sites of activation by ATP/P2X3 activation We have generated functional brain imaging (fMRI) data to suggest that the different brain circuits in receipt of nodose and jugular ganglia neuron inputs (as identified in animal studies) are conserved in humans. When inhaled, the tussigenic compound capsaicin (from hot chili peppers) indiscriminately stimulates both nodose and jugular chemosensitive afferents and we have published that capsaicin inhalation produces brain activations in the primary sensory, anterior and mid-insula, cingulate, premotor, motor and orbitofrontal cortices. These regions are presumed to encode perceptual awareness of airway irritation, and the associated emotional, cognitive and behavioral (motor) consequences. For example, activity in the human primary sensory cortex (which receives jugular ganglia inputs in animal studies) correlates with an individual's perception of airway irritation (their perceived need/ urge to cough) while activity in the insula (in receipt of nodose inputs) relates closely to the actual magnitude of the delivered stimulus independent of perception. We have now built upon these published findings by using high resolution brainstem fMRI during the inhalation of ATP (expected to only activate P2X2/3 expressing nodose-derived airway afferents) versus capsaicin (expected to activate both jugular and nodose chemosensitive afferents). Our results are striking and reveal that ATP inhalation evokes an in increased signal level in the brainstem regions corresponding to the nTS, while capsaicin inhalation produces activations in both the nTS and in an area of the dorsal spinal trigeminal nucleus on the lateral margins of the brainstem that contains the paratrigeminal nucleus. Indeed, our healthy participants did not cough as much to ATP compared to capsaicin, consistent with studies cough in animals and humans and the relatively poor cough-evoking properties of ATP in healthy humans. However, the perception of airway irritation was identical between ATP and capsaicin stimuli. We believe that cough production will ultimately be dependent upon activation of the neural circuit that integrates in the paratrigeminal nucleus (i.e.' the jugular afferent pathway) and therefore we hypothesize that there is an upregulation of the capacity of ATP to act via jugular ganglia pathways in chronic cough patients.

The fMRI studies described above provide an exciting opportunity to assess for the first time which primary airway afferent pathways are likely excited or sensitized by ATP and, in turn, what aspects of the central processing of airway sensory information is altered by ATP. We have reported previously that patients with chronic cough display functional brain responses consistent with a state of central sensitization that closely resembles the central sensitization accompanying chronic pain.

We will extend upon these findings by determining whether ATP-sensitive pathways in the brainstem and brain are altered in patients with chronic cough, and in doing so provide insight into whether ATP effects vagal afferent processing through an interaction with nodose and/ or jugular neural pathways.

ELIGIBILITY:
Inclusion Criteria:

* Patients with physician diagnosed chronic refractory cough (cough lasting >8 weeks).
* > 18 years of age
* Must be cognitively impaired

Exclusion Criteria:

* People with contraindications to MRI scanning (i.e. metal implants, claustrophobia).
* History of uncontrolled asthma or chronic respiratory disease (other than refractory cough).
* Evidence of an allergic reaction to capsaicin (chilli).
* Pregnant women.
* Smoking, current or recent history (last 6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mazzone, PhD, Principal Investigator — University of Melbourne
Locations (1):
- The University of Melbourne, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Background] Chung KF, Pavord ID. Prevalence, pathogenesis, and causes of chronic cough. Lancet. 2008 Apr 19;371(9621):1364-74. doi: 10.1016/S0140-6736(08)60595-4. PMID 18424325
- [Background] Morice AH, Jakes AD, Faruqi S, Birring SS, McGarvey L, Canning B, Smith JA, Parker SM, Chung KF, Lai K, Pavord ID, van den Berg J, Song WJ, Millqvist E, Farrell MJ, Mazzone SB, Dicpinigaitis P; Chronic Cough Registry. A worldwide survey of chronic cough: a manifestation of enhanced somatosensory response. Eur Respir J. 2014 Nov;44(5):1149-55. doi: 10.1183/09031936.00217813. Epub 2014 Sep 3. PMID 25186267
- [Background] Chung KF, McGarvey L, Mazzone SB. Chronic cough as a neuropathic disorder. Lancet Respir Med. 2013 Jul;1(5):414-22. doi: 10.1016/S2213-2600(13)70043-2. Epub 2013 May 3. PMID 24429206
- [Background] Mazzone SB, McLennan L, McGovern AE, Egan GF, Farrell MJ. Representation of capsaicin-evoked urge-to-cough in the human brain using functional magnetic resonance imaging. Am J Respir Crit Care Med. 2007 Aug 15;176(4):327-32. doi: 10.1164/rccm.200612-1856OC. Epub 2007 Jun 15. PMID 17575093
- [Background] Ando A, Smallwood D, McMahon M, Irving L, Mazzone SB, Farrell MJ. Neural correlates of cough hypersensitivity in humans: evidence for central sensitisation and dysfunctional inhibitory control. Thorax. 2016 Apr;71(4):323-9. doi: 10.1136/thoraxjnl-2015-207425. Epub 2016 Feb 9. PMID 26860344
- [Background] Abdulqawi R, Dockry R, Holt K, Layton G, McCarthy BG, Ford AP, Smith JA. P2X3 receptor antagonist (AF-219) in refractory chronic cough: a randomised, double-blind, placebo-controlled phase 2 study. Lancet. 2015 Mar 28;385(9974):1198-205. doi: 10.1016/S0140-6736(14)61255-1. Epub 2014 Nov 25. PMID 25467586

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were initially screened via telephone interviews for inclusion and exclusion criteria and gave written, informed consent prior to study enrolment. Refractory and unexplained chronic cough were diagnosed by a respiratory or laryngology specialist or general practitioner and inclusion required cough of at least 6 months duration with no abnormalities on chest X-ray or CT scan.
Groups:
- Chronic Cough Participant: Twenty-nine (29) Idiopathic chronic cough patients, defined as refractory to disease modifying therapies (eg anti-asthma medications), were recruited.
  Participants attended two sessions. In the first they inhaled in a single breath nebulized solutions of increasing doses of Adenosine Triphosphate (ATP; 0.2-300 microM) and capsaicin (0.5-125 microM) to determine their individual cough and urge-to-cough thresholds.
  In the second session, participants underwent functional brain imaging (fMRI) for 1 hour while inhaling over 24 seconds randomly administered nebulized solutions of saline, or threshold doses of ATP or capsaicin.
- Healthy Control Participant: Twenty-nine (29) appropriately age and sex matched healthy non-smoking individuals were recruited as the comparison group.
  Participants attended two sessions. In the first they inhaled in a single breath nebulized solutions of increasing doses of Adenosine Triphosphate (ATP; 0.2-300 microM) and capsaicin (0.5-125 microM) to determine their individual cough and urge-to-cough thresholds.
  In the second session, participants underwent functional brain imaging (fMRI) for 1 hour while inhaling over 24 seconds randomly administered nebulized solutions of saline, or threshold doses of ATP or capsaicin.
Period: Overall Study
Arm/Group | Chronic Cough Participant | Healthy Control Participant
Started | 29 | 29
Completed | 28 | 28
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Cough Participant | Healthy Control Participant | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (12.2) | 59.7 (12.0) | 60.1 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 10 | 10 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 29 | 29 | 58
Hull Cough Hypersensitivity Questionnaire (HARQ) score [Mean (Standard Deviation); unit: units on a scale] — Participants will be asked to self-report on symptoms related to airway reflux. Each item requires a rating on a 6-point Likert scale from 0 to 5 and is related to an aspect of airway reflux. The HARQ is scored by adding the total ratings (range 0-70). A higher score indicates a worse outcome.
  units on a scale | 33.1 (13.1) | 2.3 (2.8) | 17.5 (18.1)
Newcastle Laryngeal Hypersensitivity Questionnaire (LHQ) score [Mean (Standard Deviation); unit: units on a scale] — Participants will be asked to self-report on sensations related to laryngeal hypersensitivity. Each item requires a rating on a 7-point Likert scale from 1 to 7 and is related to an upper airway sensation in one of three domains (throat obstruction, throat pain/thermal), throat tickle). The HLQ is scored by averaging the ratings in each domain and then adding the average domain scores (range 3-21). A higher score indicates a better outcome.
  units on a scale | 14.8 (3.0) | 20.1 (1.1) | 17.5 (3.5)
Leicester Cough Questionnaire (LCQ) score [Mean (Standard Deviation); unit: units on a scale] — Participants will be asked to self-report on the impact of cough on their quality of life. Each item requires a rating on a 7-point Likert scale from 1 to 7 and is related to the impact of cough in one of three domains (physical, psychological social). The LCQ is scored by averaging the ratings in each domain and then adding the average domain scores (range 3-21). A higher score indicates a better outcome.
  units on a scale | 13.9 (3.6) | 20.8 (0.3) | 17.3 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Brainstem Neural Activations to Capsaicin
Description: fMRI will be used to determine the location and magnitude of neural responses in the brainstem during Capsaicin inhalation: in particular, the nucleus of the solitary tract and the paratrigeminal nucleus. fMRI non-invasively measures Blood Oxygen Level Dependent (BOLD) signals in the brain which can be used to identify regions of the brain that increase activity associated with the inhaled stimuli. BOLD signals detected are to be reported as % BOLD signal change in response to Capsaicin greater than control saline.
Time Frame: fMRI was performed in a single session on the day of the cough challenge testing session and not more than seven days after.
Population: Cough participants displayed characteristic signs and symptoms of refractory chronic cough. 1 participant from each group withdrew prior to completion of the primary endpoint investigation.
Measure: Mean (Standard Deviation); unit: Percentage change in BOLD signal
Groups:
- Chronic Cough Participant: Twenty-nine (29) refractory chronic cough patients, defined as refractory to disease modifying therapies (eg anti-asthma medications), were recruited.
  Participants attended two sessions. In the first they inhaled in a single breath nebulized solutions of increasing doses of Adenosine Triphosphate (ATP; 0.2-300 microM) and capsaicin (0.5-125 microM) to determine their individual cough and urge-to-cough thresholds.
  In the second session, participants underwent functional brain imaging (fMRI) for 1 hour while inhaling over 24 seconds randomly administered nebulized solutions of saline, or threshold doses of ATP or capsaicin.
Arm/Group | Chronic Cough Participant | Healthy Control Participant
Number analyzed (Participants) | 28 | 28
Percentage change in BOLD signal
  %BOLD signal Change: Nucleus of the Solitary Tract | 0.09 (0.60) | 0.39 (0.47)
  %BOLD signal Change: Paratrigeminal Nucleus | -0.14 (0.69) | 0.44 (1.06)
Statistical Analysis 1: Comparison: Chronic Cough Participant vs Healthy Control Participant; Mann-Whitney U tests for non-parametric data; Test type: Other; p = 0.0028, Wilcoxon (Mann-Whitney) — No multiple comparisons as region of interest analysis defined a priori

2. Primary Outcome: Brainstem Neural Activations to ATP
Description: fMRI will be used to determine the location and magnitude of neural responses in the brainstem during ATP inhalation: in particular, the nucleus of the solitary tract and the paratrigeminal nucleus. fMRI non-invasively measures Blood Oxygen Level Dependent (BOLD) signals in the brain which can be used to identify regions of the brain that increase activity associated with the inhaled stimuli. BOLD signals detected are to be reported as % BOLD signal change in response to ATP greater than control saline.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change in BOLD signal
Groups:
- Chronic Cough Participant: Twenty-five (25) Idiopathic chronic cough patients, defined as refractory to disease modifying therapies (eg anti-asthma medications), will be recruited.
  Participants will attend two sessions. In the first they will inhale in a single breath a nebulized solutions of increasing doses of Adenosine Triphosphate (ATP; 0.2-300 microM) and capsaicin (0.5-125 microM) to determine their individual cough and urge-to-cough thresholds. In the second session, participants will undergo functional brain imaging (fMRI) for 1 hour while inhaling over 24 seconds randomly administered nebulized solutions of saline, or threshold doses of ATP or capsaicin.
  Adenosine Triphosphate: Participants will inhale escalating concentrations of Adenosine Triphosphate (ATP) to induce cough and the urge-to-cough
  Capsaicin: Participants will inhale escalating concentrations of capsaicin to induce cough and the urge-to-cough
  Functional Brain Imaging: Participants will have scans of their brain activity using 3 Tesla (3T) brainstem restricted functional brain imaging (fMRI)
- Healthy Control Participant: Twenty-five (25) appropriately age and sex matched healthy non-smoking individuals will be recruited as the comparison group.
  Participants will attend two sessions. In the first they will inhale in a single breath a nebulized solutions of increasing doses of ATP (0.2-300 microM) and capsaicin (0.5-125 microM) to determine their individual cough and urge-to-cough thresholds. In the second session, participants will undergo fMRI for 1 hour while inhaling over 24 seconds randomly administered nebulized solutions of saline, or threshold doses of ATP or capsaicin.
  Adenosine Triphosphate: Participants will inhale escalating concentrations of Adenosine Triphosphate (ATP) to induce cough and the urge-to-cough
  Capsaicin: Participants will inhale escalating concentrations of capsaicin to induce cough and the urge-to-cough
  Functional Brain Imaging: Participants will have scans of their brain activity using 3 Tesla (3T) brainstem restricted functional brain imaging (fMRI)
Arm/Group | Chronic Cough Participant | Healthy Control Participant
Number analyzed (Participants) | 28 | 28
Percent change in BOLD signal
  %BOLD signal Change: Nucleus of the Solitary Tract | 0.04 (0.47) | 0.28 (0.58)
  %BOLD signal Change: Paratrigeminal Nucleus | 0.01 (0.65) | 0.58 (0.71)
Statistical Analysis 1: Comparison: Chronic Cough Participant vs Healthy Control Participant; Mann-Whitney U tests for non-parametric data; Test type: Other; p = 0.0070, Wilcoxon (Mann-Whitney) — No multiple comparisons as region of interest analysis defined a priori

3. Secondary Outcome: Behavioral Responses During Cough Challenge Testing: Cough Sensitivity to Capsaicin
Description: Participant responses (cough and the urge-to-cough) evoked by Capsaicin will be measured by counting audible coughs to doubling doses of Capsaicin and by asking participants to rate their perception of urge-to-cough using visual analogue scales (VAS) to each dose. Thresholds for cough sensitivity are to be reported as microM. Cu is the threshold dose required to elicit a non-zero urge-to-cough rating. C2 is the threshold dose required to elicit two audible coughs. Smax is the largest dose that could be inhaled for 24s without eliciting an audible cough. fMRI dose was the dose used during fMRI scanning.
Time Frame: Thresholds for cough sensitivity were measured during a 1 hr session prior to fMRI scanning
Population: Cough participants displayed characteristic signs and symptoms of refractory chronic cough.
Measure: Mean (Standard Error); unit: microM
Arm/Group | Chronic Cough Participant | Healthy Control Participant
Number analyzed (Participants) | 29 | 29
microM
  Capsaicin Urge to Cough threshold Cu | 0.91 (5.25) | 2.00 (2.75)
  Capsaicin Cough threshold C2 | 3.80 (4.90) | 12.89 (2.75)
  Capsaicin maximum tolerable dose Smax | 0.91 (4.27) | 3.02 (3.47)
  Capsaicin fMRI dose | 0.79 (4.17) | 1.66 (3.39)
Statistical Analysis 1: Comparison: Chronic Cough Participant vs Healthy Control Participant; Test type: Other — Group comparisons (Cough versus healthy) for each measurement using repeated measures ANOVA; p = 0.0019, ANOVA; with repeated measures

4. Secondary Outcome: Behavioral Responses During Cough Challenge Testing: Cough Sensitivity to ATP
Description: Participant responses (cough and the urge-to-cough) evoked by ATP will be measured by counting audible coughs to doubling doses of ATP and by asking participants to rate their perception of urge-to-cough using visual analogue scales (VAS) to each dose. Thresholds for cough sensitivity are to be reported as milliM. Cu is the threshold dose required to elicit a non-zero urge-to-cough rating. C2 is the threshold dose required to elicit two audible coughs. Smax is the largest dose that could be inhaled for 24s without eliciting an audible cough. fMRI dose was the dose used during fMRI scanning.
Time Frame: Thresholds for cough sensitivity were measured during a 1 hr session prior to fMRI scanning
Population: Cough participants displayed characteristic signs and symptoms of refractory chronic cough.
Measure: Mean (Standard Error); unit: milliM
Arm/Group | Chronic Cough Participant | Healthy Control Participant
Number analyzed (Participants) | 29 | 29
milliM
  ATP Urge to Cough threshold Cu | 1.29 (4.27) | 2.75 (3.63)
  ATP Cough threshold C2 | 5.75 (7.08) | 57.54 (4.79)
  ATP maximum tolerable dose Smax | 2.82 (5.75) | 19.95 (5.89)
  ATP fMRI dose | 2.82 (5.50) | 12.02 (4.47)

5. Secondary Outcome: Behavioral Responses to Cough Challenge Testing: Urge to Cough Ratings to Capsaicin and ATP
Description: Participant responses (cough and the urge-to-cough) evoked by ATP will be measured by counting audible coughs to doubling doses of ATP and by asking participants to rate their perception of urge-to-cough using visual analogue scales (VAS) to each dose.Urge-to-cough score is reported by the participant using a Bog scale ranging from 0 (no urge) to 10 (most intense urge imaginable) where the higher score, the worse the outcome. Cu is the threshold dose required to elicit a non-zero urge-to-cough rating. C2 is the threshold dose required to elicit two audible coughs. Smax is the largest dose that could be inhaled for 24s without eliciting an audible cough. fMRI dose was the dose used during fMRI scanning.
Time Frame: Urge-to-cough ratings were reported during the 1 hour cough challenge testing session and during the subsequent fMRI scanning session
Population: Cough participants displayed characteristic signs and symptoms of refractory chronic cough.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Chronic Cough Participant | Healthy Control Participant
Number analyzed (Participants) | 29 | 29
Score on a scale
  Capsaicin Urge to Cough rating at Cu | 2.07 (2.03) | 1.61 (1.47)
  Capsaicin Urge to Cough rating at C2 | 4.48 (2.32) | 6.80 (2.29)
  ATP Urge to Cough rating at Cu | 2.31 (2.12) | 1.80 (1.65)
  ATP Urge to Cough rating at C2 | 5.03 (2.57) | 6.43 (2.26)
  Capsaicin fMRI urge to cough rating | 3.65 (2.06) | 3.89 (1.97)
  ATP fMRI urge to cough rating | 2.90 (1.41) | 3.93 (2.10)
  Saline fMRI urge to cough rating | 0.86 (1.20) | 0.44 (0.71)
Statistical Analysis 1: Comparison: Chronic Cough Participant vs Healthy Control Participant; Test type: Other — Group-wise comparisons using unpaired t-tests or one way ANOVA; p < 0.0001, ANOVA

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events during the two sessions they attended: the 1 hour cough challenge testing session and subsequent 1 hour fMRI scanning session.
Groups:
- Chronic Cough Participant: Twenty-five (29) Idiopathic chronic cough patients, defined as refractory to disease modifying therapies (eg anti-asthma medications), were recruited.
  Participants attended two sessions. In the first they inhaled in a single breath a nebulized solutions of increasing doses of Adenosine Triphosphate (ATP; 0.2-300 microM) and capsaicin (0.5-125 microM) to determine their individual cough and urge-to-cough thresholds. In the second session, participants underwent functional brain imaging (fMRI) for 1 hour while inhaling over 24 seconds randomly administered nebulized solutions of saline, or threshold doses of ATP or capsaicin.
  Adenosine Triphosphate: Participants inhaled escalating concentrations of Adenosine Triphosphate (ATP) to induce cough and the urge-to-cough
  Capsaicin: Participants inhaled escalating concentrations of capsaicin to induce cough and the urge-to-cough
  Functional Brain Imaging: Participants had scans of their brain activity using 3 Tesla (3T) brainstem restricted functional brain imaging (fMRI)
- Healthy Control Participant: Twenty-five (29) appropriately age and sex matched healthy non-smoking individuals were recruited as the comparison group.
  Participants attended two sessions. In the first they inhaled in a single breath a nebulized solutions of increasing doses of ATP (0.2-300 microM) and capsaicin (0.5-125 microM) to determine their individual cough and urge-to-cough thresholds. In the second session, participants underwent fMRI for 1 hour while inhaling over 24 seconds randomly administered nebulized solutions of saline, or threshold doses of ATP or capsaicin.
  Adenosine Triphosphate: Participants inhaled escalating concentrations of Adenosine Triphosphate (ATP) to induce cough and the urge-to-cough
  Capsaicin: Participants inhaled escalating concentrations of capsaicin to induce cough and the urge-to-cough
  Functional Brain Imaging: Participants had scans of their brain activity using 3 Tesla (3T) brainstem restricted functional brain imaging (fMRI)
Arm/Group | Chronic Cough Participant | Healthy Control Participant
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT03722849/Prot_SAP_ICF_000.pdf